CLINICAL TRIAL: NCT04020666
Title: Effects of Urinary Kallidinogenase on NIHSS Score, mRS Score, and Fasting Glucose Levels in Acute Ischemic Stroke Patients With Abnormal Glucose Metabolism: a Prospective Cohort Study
Brief Title: Effects of Urinary Kallidinogenase in Acute Ischemic Stroke Patients With Abnormal Glucose Metabolism
Status: Completed | Type: Observational
Sponsor: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2016261
Record Dates: First submitted 2019-07-02; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2016-12

CONDITIONS: Acute Ischemic Stroke; Abnormal Glucose Metabolism
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- HUK group: On the basis of routine treatment for cerebral infarction, patients in the HUK group were also given Urinary Kallidinogenase at 0.15 PNA unit/day, for a 10-day course.
  Interventions: Drug: Urinary Kallidinogenase
- control group: The control group were given routine treatment for cerebral infarction, including anti-platelet aggregation, anticoagulation, lipid-lowering and plaque stabilizing, free radical scavenging, nerve nutrition and brain protection.

INTERVENTIONS:
Drug: Urinary Kallidinogenase
  Other Names: Kai Li Kang
  Groups: HUK group

SUMMARY:
Urinary kallidinogenase may assist recovery acute ischemic stroke. This study evaluated the impact of urinary kallidinogenase on NIHSS score, modified Rankin scale (mRS) score and fasting glucose levels in patients with AIS combined with diabetes mellitus and impaired fasting glucose.

DETAILED DESCRIPTION:
Patients with AIS and abnormal glucose metabolism were enrolled in this prospective cohort study and divided into two groups. The HUK group were treated with urinary kallidinogenase and standard treatment, the control group received standard treatment. NIHSS scores, mRS scores and fasting blood glucose were evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years (male or female)
* Patients were admitted to hospital within 72h of stroke onset
* Diagnosis of acute ischemic stroke according to the criteria stated in the Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke in China (2010), and patients were confirmed as acute ischemic cerebrovascular disease by head computed tomography (CT) or magnetic resonance imaging (MRI) and diffusion weighted imaging (DWI)
* NIHSS score ranged from 3-21 points
* Patients were previously diagnosed with type 2 diabetes, in which they were in line with the 2006 WHO diagnostic criteria for diabetes, or they had fasting blood glucose of 6.1-6.9mmol/L and glycosylated hemoglobin (HbA1C) of>6.1%
* Patients could cooperate with the test and evaluation of relevant indicators in the trial.

Exclusion criteria:

* Pregnant or lactating women
* Patients with severe heart, liver and kidney dysfunction
* Patients with a history of cerebrovascular disease and who still suffered from serious neurological dysfunction that had an influence on the trial
* Patients with physical disabilities, joint deformities or muscle lesions
* Patients were confirmed with intracranial hemorrhage by CT
* Patients were allergic to the study drug
* Patients suffering from severe systemic infection
* Patients who had participated in other clinical trials within 1 month
* For any reason, the researchers believed that the subject was unlikely to complete the study (such as cerebral infarction caused by cerebral embolism, intracranial arteritis, cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy (CADASIL) and moyamoya disease; patients undergoing thrombolysis or thrombectomy after admission; patients and their families were unable to cooperate with follow-up.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AIS combined with diabetes mellitus and impaired fasting glucose who was meets the Inclusion and Exclusion Criteria were enrolled in this prospective cohort study and divided into two groups.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
NIHSS Score at 90 Days | at 90 days after admission
  Comparison of NIHSS score between the control and HUK group at 90 days

SECONDARY OUTCOMES:
NIHSS Score at 10 Days、30 Days | at 10 days, 30 days after admission
  Comparison of NIHSS score between the control and HUK group at 10days、30days.
Factors related to Non-General Recovery (90-day NIHSS was reduced by <90%) | at 90 days after admission
  Based on NIHSS score，multivariate analysis was performed to evaluate the factors related to non-general recovery (90-day NIHSS was reduced by <90%) for all patients.
  Evaluation of NIHSS score: General recovery was when NIHSS score was reduced by 90%-100%; Non-general recovery referred to when NIHSS score was reduced by <90%.
mRS Score | 10 days, 30 days, and 90 days after admission
  The mRS score of 10 days after admission was taken as the baseline.Comparison of mRS score between the control and HUK group at 30days、90days.
  Based on mRS，multivariate analysis was also performed to evaluate the factors related to poor curative effect (90-day mRS ≥3) for all patients.
  Evaluation of mRS score: mRS score of 0-2 points referred to a good curative effect, and 3-5 points referred to a poor curative effect.
fasting glucose levels | at admission and 10 days after admission
  Comparison of the change in fasting glucose levels between the control and HUK group at admission and 10days.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaopeng Wang, MD, Principal Investigator — The Second Hospital of Hebei Medical University